CLINICAL TRIAL: NCT01481987
Title: Retinal Sensitivity and Optical Coherence Tomography Findings in Eyes With Idiopathic Epiretinal Membrane
Brief Title: Microperimetry and Optical Coherence Tomography (OCT) in Idiopathic Epiretinal Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Principal Investigator, Nicot Frederic, Head of research unit in Ophthalmology department, Centre Hospitalier Universitaire Dijon
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Rodica 01
Record Dates: First submitted 2011-11-21; First posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Epiretinal Membrane
Keywords: Microperimetry; OCT; idiopathic epiretinal membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epiretinal Membrane (Experimental): The investigators prospectively included 49 eyes of 49 patients with idiopathic ERM for which surgical treatment had been planned.
  Interventions: Procedure: Epiretinal Membrane Surgical treatment
- Control (No Intervention): Subjects with normal visual acuity and OCT profile

INTERVENTIONS:
Procedure: Epiretinal Membrane Surgical treatment — epiretinal membrane peeling
  Arms: Epiretinal Membrane

SUMMARY:
Purpose: To evaluate macular sensitivity and its correlation with visual acuity and Spectral Domain Optical Coherence Tomography (SD-OCT) in eyes with idiopathic epiretinal membrane (ERM).

Design: Cross sectional case-control series.

Methods:

Setting: Dijon University Hospital. Patients: Forty nine patients (49 eyes) with idiopathic ERM and twenty-seven healthy patients (27 eyes) as a control group.

Main outcome measurement: Microperimetry, Spectral Domain Optical Coherence Tomography (SD-OCT).

ELIGIBILITY:
Inclusion Criteria:

* Epiretinal Membrane

Exclusion Criteria:

* Age related macular degeneration
* Diabetic macular edema

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Macular sensitivity | 12 months
  The objective of this study was to assess macular function by measuring its sensitivity using microperimetry in patients with idiopathic ERM every three months up to one year. We compared the results of macular sensitivity to the best-corrected visual acuity (BCVA) and the OCT data to better understand the structure-function relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Creuzot-Garcher, MD, PhD, Principal Investigator — CHU Dijon
Locations (1):
- Ophthalmology Department CHU Dijon, Dijon, Burgundy, France